CLINICAL TRIAL: NCT00855244
Title: Metabolic Syndrome in Bone Marrow Transplant Survivors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator left the institution
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB09-00023
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Metabolic Syndrome
Keywords: Bone marrow transplantation
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMT survivors (Other): Diagnostic exams
  Interventions: Other: Diagnostic exams

INTERVENTIONS:
Other: Diagnostic exams — Growth hormone stimulation testing, oral glucose tolerance test, hyperinsulinemic euglycemic clamp

SUMMARY:
Life for long-term bone marrow transplant patients is complicated by endocrine late effects including growth hormone (GH) deficiency, thyroid hormone deficiency and sex steroid deficiency. Recently, studies have also identified problems with metabolic syndrome in adult bone marrow transplant (BMT) survivors. Metabolic syndrome has been identified as a constellation of insulin resistance, truncal obesity and high lipid levels (dyslipidemia) and is associated with an increased risk of type 2 diabetes and cardiovascular disease. Thus the early identification of metabolic syndrome is important. To date, studies have not identified how young an age metabolic syndrome begins in BMT survivors.

The investigators' study will consist of two aims:

1. Evaluation of children who have survived BMT for growth hormone deficiency, abnormal lipid metabolism, hypothyroidism and gonadal dysgenesis. The investigators will utilize growth hormone stimulation testing, sex steroid levels, an oral glucose tolerance test (OGTT) and fasting lipid profile to evaluate for concomitant endocrinopathy, prediabetes and impaired glucose tolerance in a cohort of BMT survivors.
2. Cross-sectional study of peripheral and hepatic insulin sensitivity in children surviving BMT using a hyperinsulinemic euglycemic clamp and the stable isotope 6,6 [2H2] glucose. These aims will provide pilot data to power the first definitive study of insulin resistance in childhood BMT survivors.

DETAILED DESCRIPTION:
Specific aim 1: Surveillance for endocrinopathy

* We will test for defects in the growth hormone (GH) axis utilizing GH stimulation testing. Briefly the patient (subject) will have studies conducted in the fasted state using two independent secretagogues (arginine and clonidine) per procedures utilized in endocrine clinical practice (See appendix for protocol). GH deficiency will be identified in those subjects whose stimulated GH value is < 10 ng/dl at all time points, according to standard criteria. We will also evaluate IGF-1 and IGFBP-3 levels and results will be interpreted per age normal values. As part of our surveillance for GH axis defects, we will obtain a bone age X-ray. Results will be interpreted according to the standards of Greulich and Pyle.
* Sex steroid levels. Testing for estrogen and testosterone levels can be done on the same day and at the same time as the GH stimulation tests. Results will be compared to bone age matched normal values as published by Esoterix Laboratory (Calabasas Hills, CA).
* OGTT- A 2-hour oral glucose tolerance test (OGTT) will be conducted at or before 9 AM, following an overnight fast. To minimize discomfort, EMLA® cream will be placed on the site for intravenous catheter (IV) insertion for 30 minutes before the IV is placed. The IV will be placed in an antecubital vein by an experienced nurse. Baseline blood samples will be withdrawn from the IV. The patient will then drink a glucola (1.75 gms CHO/kg, max 75 gms) over 3 minutes. Blood samples will be withdrawn from the IV at 30, 60 and 120 minutes following Glucola ingestion. Blood will be analyzed immediately using an YSI glucose analyzer (Yellow Springs OH) for serum glucose levels. Glucose tolerance will be categorized according to World Health Organization17. Additional blood will be collected and frozen for later analysis of insulin levels to be analyzed in the PI's laboratory.
* A fasting blood sample will be obtained for later evaluation of a fasting lipid profile. This will be conducted in the NCH laboratory. Values will be analyzed according to published age normal values18.
* We will measure waist circumference and report according to pediatric normal values6.

Specific aim 2:

* Measurement of hepatic glucose production (HGP) and protein turnover. Patients will be asked to spend the night in the Clinical Study Center (arrive by 9 p.m.). He/she will remain NPO, except for sugar- and caffeine-free liquids after 9 p.m. Prior to going to sleep, using EMLA® cream, an IV catheter will be inserted into the antecubital vein. At 4:00 a.m. we will begin infusion of stable isotopes [1-13C] NaHCO3 (bolus 0.2 mg/kg then 0.6 mg/kg/hr), [1-13C] leucine (bolus 0.35 mg/kg followed by 0.65 mg/kg/hr) and 6,6-[2H2]glucose (bolus 2.5 grams/kg followed by constant infusion of 2.0 mg/kg/hour) for 3.0 hours (isotopic equilibration period). Blood will be drawn at baseline and again after isotopic equilibration. Samples will be centrifuged and the serum frozen for future analysis by mass spectrometry in the P.I.'s laboratory. We and others have previously described these methods.20 Additionally, we will assess resting energy expenditure (REE) by 30 minute hood indirect calorimetry using the VMax calorimeter (Viasys Healthcare, Yorba Linda, CA).
* Measurement of hepatic and peripheral insulin resistance using a hyperinsulinemic euglycemic clamp. We will measure hepatic and peripheral insulin sensitivity using a hyperinsulinemic euglycemic clamp in conjunction with continued 6,6-[2H2]glucose. Again using EMLA® cream, a second IV catheter will be inserted retrograde into the back of the opposite hand and the hand will be placed in a warming box. Steady state blood will be collected from this catheter.

At 7 a.m. we will begin the clamp. Insulin will be infused initially at 10 mU/m2/min. After at least 2 hours (or longer if steady state has not occurred), the insulin infusion rate will be increased to 40 mU/m2/min. The second dose will be continued for at least 2 hours, or longer until steady-state has occurred. During insulin infusion, the patient will also receive an infusion of 20% dextrose. The rate of dextrose infusion will be adjusted every 5 - 15 minutes to keep plasma glucose 88-95 mg/dl. Plasma glucose will be measured every 5-10 minutes at bedside using an automated glucose oxidase technique (Glucose Analyzer; YSI, Yellow Springs, OH). To prevent hypokalemia and hypophosphatemia, K2HPO4 will be infused throughout the study, and serum potassium levels will be measured at baseline and at the end of the study. Blood will be collected for later detection of 6H6 in plasma before infusion of isotope (baseline), at steady state (just before insulin infusion) and at the end of each insulin infusion "step." We will also collect blood for analysis of plasma insulin levels at these time points. Our group has previously reported the details of these methods21.

Peripheral insulin sensitivity will be reported as half maximal glucose disposal rate (in milligrams/kilogram/minute) according to the amount of glucose required to maintain serum glucose levels 88-93 mg/dl, at an insulin dose of 40 mU/m2/min. This will be taken as the mean of three 15-minute intervals once steady-state has been achieved. Hepatic insulin sensitivity will be quantified by comparing HGP at baseline to HGP as measured at the end of the 10mU/m2/min clamp.

We will measure bone density using a DXA scan (Lunar Prodigy) which will include measure of whole body, hip and spine for both bone mineral density and content. Measurements will be compared to age- and gender- matched normals and converted to Z scores (www.bcm.edu/bodycomplab).

**Safety issues: We have previously used the hyperinsulinemic euglycemic clamp in over 200 adults and in 6 adolescents. At no time have any of our subjects experienced hypoglycemia. We reduce risk by measuring the glucose level at bedside every 5 -15 minutes and adjusting the dextrose infusion within one minute of measuring plasma glucose. The P.I. is present at each and every clamp procedure and uses the same skilled nurse as an assistant. This will be the case for studies done at any site. We are using the minimal model as modified for children, which greatly minimizes the loss of blood. The maximum blood loss for participation in this study is estimated to be 52 cc's per child. The stable isotope methods have been used extensively in both pregnant women and in children.

In Vitro Methods:

* Determination of isotope enrichment- 6H6-enrichment of plasma will be measured following derivatization using a Hewlett Packard 5989A gas chromatograph/mass spectrometer in the electron impact mode. Measures will be conducted in the applicant's laboratory.
* Hormone and other analysis- Insulin and C-peptide levels will be measured using a doubly labeled antibody technique in the applicant's laboratory. Hemoglobin A1c and fasting lipid profiles will be measured by the laboratory at Nationwide Children's Hospital.

ELIGIBILITY:
Inclusion Criteria:

* One year post BMT in autogenic transplanted patients and two years from BMT in allogenic transplanted patients
* The participants may be from any ethnic group and of either gender
* Free of the following chronic medical illness (diseases possibly associated with glucose intolerance or altered insulin sensitivity): type 1 DM, HIV, chronic liver disease, cystic fibrosis, chronic renal failure, known genetic syndrome.

Exclusion Criteria:

* On-going graft vs. host disease
* Use of Megace® or another progestational agent
* Use of anabolic steroids
* Diagnosis of one of the chronic diseases listed above

Ages: 9 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2009-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
This information will be used to conduct a power analysis (Norton Power Software or NQuery Advisor) for design of a larger study. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Termuhlen, MD, Study Director — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Meacham L. Endocrine late effects of childhood cancer therapy. Curr Probl Pediatr Adolesc Health Care. 2003 Aug;33(7):217-42. doi: 10.1016/s1538-5442(03)00053-1. No abstract available. PMID 12902974
- [Background] Oberfield SE, Sklar CA. Endocrine sequelae in survivors of childhood cancer. Adolesc Med. 2002 Feb;13(1):161-9, viii. PMID 11841962
- [Background] Taskinen M, Lipsanen-Nyman M, Tiitinen A, Hovi L, Saarinen-Pihkala UM. Insufficient growth hormone secretion is associated with metabolic syndrome after allogeneic stem cell transplantation in childhood. J Pediatr Hematol Oncol. 2007 Aug;29(8):529-34. doi: 10.1097/MPH.0b013e3180f61b67. PMID 17762493